CLINICAL TRIAL: NCT07218081
Title: Cognitive Brain Aging Reversal From Deep Brain Stimulation for Alzheimer's Dementia: a Clinical Trial.
Brief Title: A Trial to Test Intermittent Deep Brain Stimulation of Nucleus Basalis of Meynert to Treat Alzheimers.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, David Blake, Professor David T. Blake, Augusta University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2300118-2
Record Dates: First submitted 2025-09-29; First posted 2025-10-20 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Alzheimer Dementia (AD)
Keywords: deep brain stimulation; alzheimer's; nucleus basalis of Meynert
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Six subjects will receive open label intermittent deep brain stimulation of the nucleus basalis of Meynert for 50 minutes daily. Six control subjects will document expected progression under normal standard of care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Intermittent deep brain stimulation of the nucleus basalis of Meynert (Experimental): Subjects will receive intermittent deep brain stimulation of the nucleus basalis of Meynert for 50 minutes each day. Assessments will be performed at onset, after four weeks of intervention, and each six months through two years.
  Interventions: Device: Intermittent deep brain stimulation of the nucleus basalis of Meynert
- Control group (No Intervention): Subjects will have matching eligility criteria as those in the experimental arm, but will receive no intervention. Assessments will be performed at study onset, and each six months through two years after onset.

INTERVENTIONS:
Device: Intermittent deep brain stimulation of the nucleus basalis of Meynert — Subjects will receive intermittent deep brain stimulation of the nucleus basalis of Meynert for 50 minutes each day.
  Arms: Intermittent deep brain stimulation of the nucleus basalis of Meynert

SUMMARY:
The purpose of this study is to test a new procedure to treat Alzheimer's disease. The procedure is called intermittent Deep Brain Stimulation (DBS) of the nucleus basalis of Meynert. There will be up to six participants enrolled at Wellstar MCG Memory Clinic. There will be another six participants similarly enrolled to act as a control group that does not receive DBS. This second group will document the course of progression of Alzheimer's disease under the normal standard of care. The main goal of the study is to determine if DBS can sustain or improve cognition in Alzheimer's disease for at least two years. Participant data, with identifying information removed, may be shared with online repositories for comparison with trials with similar subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age:65 minimum

  * Age:85 maximum
  * Probable, early-stage Alzheimer's Disease, as defined by NIA-AA 2018 criteria and positive PET for beta amyloid,
  * no Lewy-Body-dementia or other form of dementia
  * Clinical Dementia Rating (CDR) global score of 0.5-1.0 with a CBR-sb score from 2 to 6.
  * MMSE ≥ 21
  * stable psychopharmacological medication equivalent to 10 mg/day donepezil or less for at least 60 days
  * valid informed consent
  * an available caregiver willing to participate
  * subject is living at home and likely to remain at home for the study duration
  * Geriatric Depression Scale of 5 or less
  * Columbia Suicide Severity Rating Scale "No" on questions 3 through 5
  * Neuropsychiatric Inventory (NPI-Q) under 2 on 'Delusions', 'Hallucinations' or 'Agitation/Aggression' subscales

Exclusion Criteria:

* • clinical co-morbidity interfering with study (e.g. head trauma requiring medical treatment in the 2 years prior, brain tumor, subdural hematoma, or other clinically significant space-occupying lesion on brain CT or MRI), or other implant precluding high field MRI scans.

  * current major psychiatric disorder such as schizophrenia, bipolar disorder or major depressive disorder based on psychiatric consult at screening visit, or past medical history prior suicidal attempts or suicidal crises
  * Another concurrent CNS condition (ie, stroke, Parkinson's disease, Lewy-Body dementia or other form of dementia, other evidence of significant structural brain pathology).
  * Medical history of seizure disorder including epilepsy
  * Terminal illness associated with expected survival of <30 months
  * Subjects with one of these other forms of dementia in the DSM-5 heading of Neurocognitive Disorders: Lewy body disease, Frontotemporal lobar degeneration, Vascular disease, Traumatic brain injury, HIV infection, Prion disease, Parkinson's disease, Huntington's disease, or due to multiple etiologies
  * Subjects with unstable medical and neurological conditions at the discretion of the Principle Investigator

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-11-01 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Dementia Rating Scales | Two years after intervention onset
  Subjects will be evaluated using the Clinical Dementia Rating Sum of Boxes scale. The investigators seeks for half of the intervention arm participants to have better (lower) or equal scale scores two years after intervention onset than they had at onset. This scale ranges from 0 to 18, and subjects will score from 2 to 6 at study entry.
Alzheimer's Disease Assessment Scale, Cognitive Subscale | Two years of intervention
  The investigators seeks for scores on the Alzheimer's Disease Assessment Scale, Cognitive Subscale, to be equal or lower in half of the participants two years after the intervention begins compared to their value at study onset. This scale ranges from 0 to 85, and subjects at onset will likely have scores between 13 and 30.

SECONDARY OUTCOMES:
PET scans for beta amyloid | Two years after study onset.
  PET scans will be obtained at onset and annually through two years. The investigators seek for a reduction in the Standard Uptake Volume Ratio (SUVr) in the intervention arm compared to the control arm. SUVr is a ratio of image intensity in a reference region of the brain compared to the cerebral cortex. SUVr averages 1.22 in subjects diagnosed with Alzheimer's, and 1.0 in non-Alzheimer's controls.
Anxiety scales | Two years of intervention
  Subjects will receive a GAD-7 questionnaire at the same times as cognitive assessments. The investigators seek for reductions in the GAD-7 values in the intervention arm compared to the control arm. The GAD-7 scale ranges from 0 to 21, and higher scores indicate more anxiety.
Beta amyloid PET imaging, Centiloid scale. | Two years of intervention
  PET scans will be obtained from particpants at onset and annually through two years. The investigators seek for a reduction in the Centiloid Scale in the intervention arm compared to the control arm. The Centiloid scale is 0CL on average in a 45 year old normal, and 100CL in a person with Alzheimer's dementia.
PHQ-9 questionaire | Two years of intervention
  Participants will receive a PHQ-9 questionnaire at the same times as cognitive assessments. The investigators seek for reductions in this scale in the intervention arm compared to the control arm. The PHQ-9 depression scale has scores from 0 to 27, and higher scores indicate more depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Wellstar MCG Hospital, Neurology Memory Clinic, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Subject data will be de-identified. Assessment outcomes and imaging results will be uploaded to open access websites for sharing such data like ADNI.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be shared upon publication and will be available indefinitely.
Access Criteria: Access will be open.

REFERENCES:
- [Background] Sasikumar S, Cohn M, Youm A, Duncan K, Boogers A, Strafella AP, Blake DT, Fasano A. Rethinking NBM DBS: Intermittent stimulation improves sustained attention in Parkinson's disease. Brain Stimul. 2023 Nov-Dec;16(6):1643-1645. doi: 10.1016/j.brs.2023.10.014. Epub 2023 Nov 5. No abstract available. PMID 37935282
- [Background] Kumro J, Tripathi A, Lei Y, Sword J, Callahan P, Terry A, Lu XY, Kirov SA, Pillai A, Blake DT. Chronic basal forebrain activation improves spatial memory, boosts neurotrophin receptor expression, and lowers BACE1 and Abeta42 levels in the cerebral cortex in mice. Cereb Cortex. 2023 Jun 8;33(12):7627-7641. doi: 10.1093/cercor/bhad066. PMID 36939283
- [Background] Pennington KR, Debs L, Chung S, Bava J, Garin CM, Vale FL, Bick SK, Englot DJ, Terry AV Jr, Constantinidis C, Blake DT. Basal forebrain activation improves working memory in senescent monkeys. Brain Stimul. 2025 Mar-Apr;18(2):185-194. doi: 10.1016/j.brs.2025.02.002. Epub 2025 Feb 7. PMID 39924100
- [Background] Liu R, Crawford J, Callahan PM, Terry AV Jr, Constantinidis C, Blake DT. Intermittent Stimulation of the Nucleus Basalis of Meynert Improves Working Memory in Adult Monkeys. Curr Biol. 2017 Sep 11;27(17):2640-2646.e4. doi: 10.1016/j.cub.2017.07.021. Epub 2017 Aug 17. PMID 28823679